CLINICAL TRIAL: NCT06948526
Title: Clinical and Radiographic Evaluation of Moringa Oleifera Leaf Extract Versus Sodium Hypochlorite as Intracanal Irrigations in Pulpectomy of Nonvital Primary Molars: A Randomized Clinical Trial
Brief Title: Evaluation of Moringa Oleifera Leaf Extract Versus Sodium Hypochlorite in Pulpectomy of Nonvital Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lama Hatem Fouad Sobhi, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRE - Moringa Vs NaOCl
Record Dates: First submitted 2025-04-18; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Nonvital Primary Molars

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moringa Oleifera Leaf Extract Irrigation (Experimental): Participants in this arm will receive pulpectomy treatment using Moringa Oleifera leaf extract as the intracanal irrigant. The extract will be used to irrigate the root canals after working length determination, using a 3 ml syringe with a side-vented needle to minimize the risk of apical extrusion. Mechanical preparation will follow using a rotary system, and the canals will be obturated with Metapex and restored with stainless steel crowns.
  Interventions: Drug: Moringa Oleifera Leaf Extract
- Sodium Hypochlorite Irrigation (Active Comparator): Participants in this arm will receive pulpectomy treatment using 1% Sodium Hypochlorite as the intracanal irrigant. The irrigant will be applied in the same manner as in the experimental group, using a 3 ml syringe and side-vented needle following root canal instrumentation. Mechanical preparation, obturation with Metapex, and stainless steel crown placement will be performed identically to the experimental group.
  Interventions: Drug: Sodium Hypochlorite 1%

INTERVENTIONS:
Drug: Moringa Oleifera Leaf Extract — A plant-based extract derived from Moringa Oleifera leaves, used as an intracanal irrigant during pulpectomy procedures in primary molars. It is administered using a 3 ml syringe with a side-vented needle following canal preparation and working length determination. This intervention aims to evaluate the clinical and radiographic efficacy of a natural, biocompatible alternative to conventional chemical irrigants.
  Other Names: Moringa extract; Natural intracanal irrigant
  Arms: Moringa Oleifera Leaf Extract Irrigation
Drug: Sodium Hypochlorite 1% — A 1% concentration of Sodium Hypochlorite solution used as a standard intracanal irrigant in pediatric endodontics. It is administered using a 3 ml syringe with a side-vented needle after canal instrumentation. Known for its strong antimicrobial and tissue-dissolving properties, Sodium Hypochlorite serves as the active comparator in this study.
  Other Names: NaOCl; Standard chemical irrigant
  Arms: Sodium Hypochlorite Irrigation

SUMMARY:
This randomized clinical trial aims to compare the clinical and radiographic success of Moringa Oleifera leaf extract with Sodium Hypochlorite as intracanal irrigants in pulpectomy of nonvital primary molars in children aged 3-7 years. The study evaluates both clinical parameters (pain, swelling, mobility) and radiographic healing (periapical changes, root resorption) over 12 months.

DETAILED DESCRIPTION:
Effective disinfection during pulpectomy of primary molars is essential for treatment success. Sodium hypochlorite is the gold standard intracanal irrigant but presents concerns regarding cytotoxicity and taste. Moringa Oleifera, a natural agent with antimicrobial, antioxidant, and anti-inflammatory properties, may offer a biocompatible alternative. This study is a parallel-design, randomized clinical trial evaluating 50 teeth in children aged 3-7 years. Patients will be randomly allocated to either 1% Sodium Hypochlorite or Moringa Oleifera leaf extract for intracanal irrigation. Clinical and radiographic outcomes will be assessed at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Cooperative children aged between 3-7 years
* Males/Females.
* Primary molars necessitating pulpectomy diagnosed with deep dental caries with pulp necrosis and periapical pathosis or both.
* Systemically healthy children

Exclusion Criteria:

* Medically compromised and uncooperative children
* Tooth indicated for extraction due to root resorption more than two thirds of the root, teeth near exfoliation, deep subgingival caries hindering proper coronal seal.
* Mobile teeth (Miller's Grade 2 or more)
* Previous pulp therapy

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 3, 6, 12 months
  Postoperative pain will be assessed using the Visual Analog Scale (VAS), a 10-point scale where 0 represents "no pain" and 10 represents "worst possible pain." Higher scores indicate worse pain outcomes. Pain levels will be recorded at 3, 6, and 12 months post-treatment.
Soft Tissue Healing | 3, 6, 12 months
  Visual and palpation-based assessment for swelling, sinus tract, or redness.
Pain on Percussion & Mobility | 3, 6, 12 months
  Tested clinically for tenderness and abnormal mobility.

SECONDARY OUTCOMES:
Periapical Radiographic Changes | 6 and 12 months
  Evaluated using digital radiographs.
Internal/External Root Resorption | 6 and 12 months
  Identified via radiographic analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, El-Manial, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
The data will be securely stored and only accessible by the research team for analysis.

REFERENCES:
- [Background] Peretz B, Yakir O, Fuks AB. Follow up after root canal treatment of young permanent molars. J Clin Pediatr Dent. 1997 Spring;21(3):237-40. PMID 9484133
- [Background] Alharbi AM, Alharbi TM, Alqahtani MS, Elfasakhany FM, Afifi IK, Rajeh MT, Fattouh M, Kenawi LMM. A Comparative Evaluation of Antibacterial Efficacy of Moringa oleifera Leaf Extract, Octenidine Dihydrochloride, and Sodium Hypochlorite as Intracanal Irrigants against Enterococcus faecalis: An In Vitro Study. Int J Dent. 2023 Mar 14;2023:7690497. doi: 10.1155/2023/7690497. eCollection 2023. PMID 36960331